CLINICAL TRIAL: NCT05638763
Title: Cytochrome P450 Inhibition With Ketoconazole to Decrease Dosage and Costs of Dasatinib for Chronic Myelogenous Leukemia
Brief Title: Cytochrome P450 Inhibition to Decrease Dosage of Dasatinib for Chronic Myelogenous Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Fernando De la Garza Salazar (Unknown)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Department, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE22-00031
Record Dates: First submitted 2022-11-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dasatinib and ketoconazole (Experimental): Patients will receive dasatinib at a dose of 25mg orally daily for one year and ketoconazole 200mg orally two times per day for one year.
  Interventions: Drug: Dasatinib Pill; Drug: Ketoconazole Pill

INTERVENTIONS:
Drug: Dasatinib Pill — Patients will receive half pill of dasatinib 50mg (25mg/day, orally) for one year
  Other Names: Sprycel
Drug: Ketoconazole Pill — Patients will receive ketoconazole 200mg two times a day, orally, for one year.
  Other Names: Nizoral

SUMMARY:
This phase 2 single-arm study aims to demonstrate the efficacy of strong cytochrome inhibition with ketoconazole to reduce dasatinib dosage for adults with chronic myelogenous leukemia. Researchers will describe response rates and adverse events.

DETAILED DESCRIPTION:
Dasatinib is a second-generation tyrosine kinase inhibitor that is metabolized by the cytochrome P450. Dasatinib has shown efficacy in patients with chronic myelogenous leukemia. Standard-dose dasatinib is 50mg-140mg/day orally, continuously. However, when combined with a strong CYP3A4 inhibitor, a dose reduction of 75% is warranted.

This phase 2 single-arm study aims to demonstrate the efficacy of strong cytochrome inhibition with ketoconazole to reduce the dosage and costs of dasatinib for adults with chronic myelogenous leukemia. Researchers will describe cytogenetic and molecular response rates at 3, 6, and 12 months and adverse events (i.e., pleural effusion) associated with this strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Chronic myeloid leukemia in chronic phase according to the World Health Organization 2016
3. Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

1. Chronic heart disease (NYHA III-IV)
2. Bleeding disorders not attributed to the hematological malignancy
3. Pregnancy
4. Lactation
5. Chronic myeloid leukemia in blast phase
6. Organic dysfunction (Marshall score ≥2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The rate of Complete Cytogenetic Response | Up to 6 months
  B-cell antigen receptor(BCR)/Tyrosine-protein kinase-ABL1(ABL1) IS <=1% at 6 months

SECONDARY OUTCOMES:
The rate of Molecular Response (MR4) | Up to 6 months
  Log reduction in BCR/ABL of 4
The rate of Molecular Response (MR4.5) | Up to 6 months
  Log reduction in BCR/ABL of 4.5
The rate of sustained Molecular Response (MR4.5) | Up to 12 months
  Log reduction in BCR/ABL of 4.5
The proportion of non hematological side effects | Up to 12 months
  Proportion of patients that presented non hematological side effects to the intervention
The rate of Complete Cytogenetic Response | Up to 12 months
  BCR/ABL IS <=1% at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hochhaus A, Saussele S, Rosti G, Mahon FX, Janssen JJWM, Hjorth-Hansen H, Richter J, Buske C; ESMO Guidelines Committee. Chronic myeloid leukaemia: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv41-iv51. doi: 10.1093/annonc/mdx219. No abstract available. PMID 28881915
- [Background] Johnson FM, Agrawal S, Burris H, Rosen L, Dhillon N, Hong D, Blackwood-Chirchir A, Luo FR, Sy O, Kaul S, Chiappori AA. Phase 1 pharmacokinetic and drug-interaction study of dasatinib in patients with advanced solid tumors. Cancer. 2010 Mar 15;116(6):1582-91. doi: 10.1002/cncr.24927. PMID 20108303
- [Background] Naqvi K, Jabbour E, Skinner J, Anderson K, Dellasala S, Yilmaz M, Ferrajoli A, Bose P, Thompson P, Alvarado Y, Jain N, Takahashi K, Burger J, Estrov Z, Borthakur G, Pemmaraju N, Paul S, Cortes J, Kantarjian HM. Long-term follow-up of lower dose dasatinib (50 mg daily) as frontline therapy in newly diagnosed chronic-phase chronic myeloid leukemia. Cancer. 2020 Jan 1;126(1):67-75. doi: 10.1002/cncr.32504. Epub 2019 Sep 25. PMID 31553487